CLINICAL TRIAL: NCT04058834
Title: A First Human Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of Single Doses of NNC0385-0434 in Healthy Subjects and Patients With Hypercholesterolaemia
Brief Title: A Research Study Investigating How NNC0385-0434 is Tolerated in People With or Without High Cholesterol Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6434-4493; U1111-1231-4690 (Other: World Health Organization (WHO)); 2019-001746-18 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers; Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Four (4) cohorts are planned. In 3 cohorts, healthy subjects will be randomised in a 3:1 manner to receive either: 1) NNC0385-0434 or 2) Placebo (NNC0385-0434). Each cohort will last 10 weeks and there will be 3 weeks between cohorts. Following safety observation, a fourth cohort will be initiated with patients with hypercholesterolaemia. Patients will be randomised in a 2:1 manner to receive either: 1) NNC0385-0434 or 2) Placebo (NNC0385-0434).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0385-0434 (Experimental): Healthy volunteers will be randomised to one of three cohorts. In each cohort of 8 participants, 6 will receive active drug and 2 will receive placebo. Following safety observation, patients with hypercholesterolaemia will enter a fourth cohort. There will be 15 participants in this cohort.
  Interventions: Drug: NNC0385-0434
- Placebo (NNC0385-0434) (Placebo Comparator): Healthy volunteers will be randomised to one of three cohorts. In each cohort of 8 participants, 6 will receive active drug and 2 will receive placebo.
  Interventions: Drug: Placebo (NNC0385-0434)

INTERVENTIONS:
Drug: NNC0385-0434 — Healthy volunteers and patients will receive one injection s.c. (subcutaneously, under the skin)
  Arms: NNC0385-0434
Drug: Placebo (NNC0385-0434) — Healthy volunteers will receive one injection s.c.
  Arms: Placebo (NNC0385-0434)

SUMMARY:
In this study, there are two study medicines: NNC0385-0434 (the new medicine being tested) and placebo (a 'dummy' medicine). Participants will only get one of these medicines - which one is decided by chance. The study medicine for each person is chosen by a computer. A dummy medicine (placebo) looks like the study medicine but has no effect on the body. The dummy medicine needs to be used in the study to find out if the study medicine works as expected. The dose of the study medicines that participants receive will depend on which group they get into. The study has 4 groups of 8-15 participants in each. Each group will get a different dose of NNC0385-0434 or placebo. Participants and the study doctor will not know which of the study medicine/dose participants will get. However, if a participant's safety is at risk, the study doctor will be told in order to decide the future treatment. NNC0385-0434 may help to clear cholesterol from the blood. When there is less cholesterol circulating in the blood over a long period of time, then there is less risk of arteries (blood vessels) being clogged or developing diseases of the heart and blood vessels. Each participant will get one injection under the skin and will be in the study for about 4 months.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Body mass index between 20.0 kg/m^2 and 35.0 kg/m^2 (both inclusive).
* Male subjects.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.

Patients with hypercholesterolaemia:

* Body mass index between 20.0 kg/m^2 and 35.0 kg/m^2 (both inclusive).
* Male subjects.
* Aged 18-70 years (both inclusive) at the time of signing informed consent.
* Stable treatment with high- or moderate-intensity statin defined as total daily dose level of rosuvastatin equal to or above 10 mg, atorvastatin equal to or above 10 mg, simvastatin equal to or above 20 mg, pravastatin equal to or above 40 mg, lovastatin equal to or above 40 mg, fluvastatin equal to or above 80 mg, or pitavastatin equal to or above 1 mg for at least 30 days prior to enrolment and expected to remain on this dose for the remainder of the trial.

Exclusion Criteria:

Healthy volunteers:

* Male subjects who are not surgically sterilised (vasectomy) and are sexually active with female partner(s) and not using condom with spermicide combined with an effective method of contraception for their female partner(s) in the period from randomisation visit (V2) until 10 weeks following administration of the investigational medical product.
* Any disorder which in the Investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.

Patients with hypercholesterolaemia:

* Male subjects who are not surgically sterilised (vasectomy) and are sexually active with female partner(s) and not using condom with spermicide combined with an effective method of contraception for their female partner(s) in the period from randomisation visit (V2) until 10 weeks following administration of the investigational medical product.
* Any disorder which in the Investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.
* Current treatment with ezetimibe unless treatment has been with a stable dose for at least 30 days prior to enrolment and expected to remain on this dose for the remainder of the study.
* History (as declared by the subject or reported in the medical records) of heart failure or clinically significant cardiac arrhythmia.
* History (as declared by the subject or reported in the medical records) of myocardial infarction, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, peripheral vascular or cerebrovascular disease within 12 months prior to enrolment
* Planned surgery or revascularization at time of screening.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From time of first dosing (Day 1) to completion of the post-treatment follow-up visit (Day 70)
  Count

SECONDARY OUTCOMES:
AUC0-∞,0434,SD; the area under the NNC0385-0434 plasma concentration-time curve from time 0 to infinity after a single dose of s.c. NNC0385-0434 | From day of dose (Day 1) until end of treatment (Day 70)
  nmol/L*h
Cmax,0434,SD; the maximum plasma concentration of NNC0385-0434 after a single dose of s.c. NNC0385-0434 | From day of dose (Day 1) until end of treatment (Day 70)
  nmol/L
t½,0434,SD; the terminal half-life of NNC0385-0434 after a single dose of s.c. NNC0385-0434 | From time of first dosing (Day 1) to completion of the post-treatment follow-up visit (Day 70)
  h
tmax,0434,SD; the time to maximum plasma concentration of NNC0385-0434 after a single dose of s.c. NNC0385-0434 | From time of first dosing (Day 1) to completion of the post-treatment follow-up visit (Day 70)
  h
Change in fasting LDL-C levels after a single dose of s.c. NNC0385-0434 | Day 1, day 70
  Ratio to pre-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com